CLINICAL TRIAL: NCT00549029
Title: Association Analysis Between Single Nucleotide Polymorphisms in Statin-Related Genes and The Incidence of Myopathy Among Statin-Treated Patients
Brief Title: The Association of Genetic Polymorphisms With Statin-Induced Myopathy.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 200708077R
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Rhabdomyolysis; Myopathy
Keywords: muscle disorder; statins; creatine kinase
MeSH Terms: conditions — Rhabdomyolysis; Muscular Diseases | interventions — DNA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1,2: Group 1 for the patients with rhabdomyolysis Group 2 for the control without any myopathy
  Interventions: Genetic: DNA

INTERVENTIONS:
Genetic: DNA — withdraw 5~10mL blood from vein only once during the whole design

SUMMARY:
To observe not only the distribution of single nucleotide polymorphism in genes related with pharmacodynamic and pharmacokinetics alteration of statins but also to analyze the correlation between these SNPs and the incidence of statins-induced myopathy.

DETAILED DESCRIPTION:
Statins are widely prescribed for the patients with hypercholesterolemia.

Though their efficacy in preventing cardiovascular events has been shown by a large number of clinical trials, myotoxic side effects including myopathy or even more severe,rhabdomyolysis are associated with the use of statins.

Because the incidence of myopathy is various among individuals,polymorphism in genes is supposed to be the main factor.

Due to single nucleotide polymorphism in related genes,level of uptake, clearance and metabolism of statins can be seriously different among individuals resulting in various occurrence of myopathy.

Therefore, analytical study in association between SNP of statins-related genes and the incidence of myopathy is such a critical research which can be applied into clinical fields.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Rhabdomyolysis because of prescription with statins

Exclusion Criteria:

* Carnitine palmityl transferase ll deficiency
* McArdle disease
* Myoadenylate deaminase deficiency

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: National Taiwan University Hospital
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2007-08; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
genotype of specific genes | one day

SECONDARY OUTCOMES:
single nucleotide polymorphism | one day

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Hui Chen, PhD, Study Director — National Taiwan Univesity College of Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Jisun Oh, et al. Genetic determinants of statin intolerance. Lipid in Health and Disease 2007;6(7). Wei Zhang, et al. Role of BCRP 421C>A polymorphism on rosuvastatin pharmacokinetics in healthy Chinese males. Clinica Chimica Acta 2006;373:99-103. Mikko Niemi, et al. Association of genetic polymorphism in ABCC2 with hepatic multidrug resistance-associated protein 2 expression and pravastatin pharmacokinetics. Pharmacogenetics and Genomics 2006;16:801-808. Andre' BM, et al. Association of polymorphism in the cytochrome CYP2D6 and the efficacy and tolerability of simvastatin. Clin Pharmacol Ther 2001;70:546-551. K. Morimoto, et al. OATP-C(OATPO1B1)15 IS ASSOCIATED WITH LESTEROLEMIC PATIENTS. CLINICAL PHARMACOLOGY THERAPEUTICS 2005;77(2). K. Morimoto, et al. CANDIDATE OF GENETIC MARKERS FOR STATIN-INDUCED MYOPATHY IN JAPANESE PATIENTS WITH HYPERCHOLESTEROLEMIA. Drug Metabolism Reviews 2005;37(4):345.